CLINICAL TRIAL: NCT02586493
Title: An Open-label Study of the Correct Use and Ease of Use of Placebo ELLIPTA Dry Powder Inhaler in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Ease of Use and Correct Use Study of Placebo ELLIPTA® Inhaler in COPD Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201071
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Placebo; ELLIPTA inhaler; Correct use; COPD; Ease of use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo ELLIPTA inhaler (Experimental): Subjects will be provided the ELLIPTA inhaler, which is a molded plastic two-sided inhaler that holds two individual blister strips containing either lactose or a blend of lactose and magnesium stearate. Subjects will continue to use regular COPD medications throughout the study as per protocol.
  Interventions: Drug: Placebo; Other: Questionnaire

INTERVENTIONS:
Drug: Placebo — Subjects will receive 1 inhalation once-daily until visit 2.
Other: Questionnaire — ELLIPTA Inhaler Ease of Use Questionnaire is a four-point Likert scale. This questionnaire will be filled by investigator (designee) based on responses received from subject. Responses for the questionnaire are Very difficult, Difficult, Easy, Very easy. Subjects will be give either version A or B at Visit 2.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a preventable and treatable disease characterized by airflow limitation that is not fully reversible. The mainstay for treatment involves the use of inhaled medications, including short and/or long-acting bronchodilators along with inhaled corticosteroids. For inhaled medications, the choice of inhalation device is an important consideration because an inadequate technique reduces the effects of inhalation. Therefore, the development of an easy-to-use inhaler that delivers the drug to the lungs effectively, is important. This study will assess the correct use of the ELLIPTA inhaler by subjects with COPD and to assess ease of use of the ELLIPTA inhaler, as rated by those subjects determined to be using the inhaler correctly. Study will be divided into two visits i.e. Screening/Visit 1 (day 1) and Visit 2 (Day 28 +/-2) with a phone call on Day 8+/-2 days of Visit 1 to assess safety. In this multi-center, single-arm, randomised (to receive one of two versions of the ELLIPTA inhaler Ease of Use questionnaires), open-label, placebo study, only subjects who are have never used the ELLIPTA inhaler before and have an established diagnosis of COPD and receiving COPD therapy and are able to demonstrate correct use of the ELLIPTA inhaler at Visit 1 will be considered eligible to participate in this study. Approximately 252 subjects will be screened with an expectation of 208 subjects completing the study while demonstrating correct ELLIPTA inhaler use at visit 2.

ELLIPTA is a registered trademark of the GlaxoSmithKline Group of Companies.

ELIGIBILITY:
Inclusion Criteria:

* Age: >=40 years of age at Visit 1
* Diagnosis of COPD with a documented history of COPD for at least one year, in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Severity of Disease: Post albuterol/salbutamol forced expiratory volume in one second (FEV1)/ forced vital capacity (FVC) ratio <0.70 and FEV1 <=70% of predicted obtained within two years of Visit 1.
* Smoking History: Current or former (defined as subjects who have quit smoking for at least 3 months prior to Screening/Visit 1) cigarette smokers with a >10 pack-year smoking history (Number of pack years = [number of cigarettes per day divided by 20] x number of years smoked [e.g., 10 pack-years is equal to 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years]).
* Current COPD Therapy: Currently receiving maintenance (with one or more long-acting bronchodilators, such as a long-acting muscarinic antagonist (LAMA; also known as a long-acting anti-cholinergic) or long-acting beta 2-agonist (LABA) inhaler therapy (with no prior or ongoing use of ELLIPTA inhaler) for the treatment of COPD. Subjects must be able to continue using their currently prescribed COPD maintenance inhaler therapy throughout the study and as needed short acting beta-adrenergic agonist (SABA) for rescue use.
* Ability to Use Inhalers: Subject must be able to demonstrate correct use of ELLIPTA inhaler within three attempts at Visit 1.
* Males
* Females who are not pregnant or not planning a pregnancy during the study or not lactating.
* Informed Consent: Capable of giving signed and dated written informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.
* Subject understands and is willing, able, and likely to comply with study procedures and restrictions.
* Subject must be able to read, comprehend, and record information in English.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply

* Asthma: Subjects with a current primary diagnosis of asthma.
* COPD medications: Receiving only inhaled short-acting beta-adrenergic agonists, i.e., albuterol as their daily COPD therapy (as needed [prn] or regularly scheduled); Has changed maintenance COPD treatment within 4 weeks prior to Screening/Visit 1 or plans to change COPD treatment within 4 weeks of Visit 1.
* COPD/Exacerbations/Hospitalization: Subjects that have experienced a COPD exacerbation requiring systemic corticosteroids (oral, parenteral or depot) and/or antibiotics within four weeks of Visit 1. A subject must not have had any hospitalization for COPD within three months prior to Visit 1; Subjects with uncontrolled COPD, in the investigator's judgment that would affect subject's ability to evaluate "ease of use and correct use".
* Other Respiratory Disorders: Subjects with other respiratory disorders, including active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening/Visit 1.
* Oxygen: Use of long-term oxygen therapy (LTOT; defined as oxygen therapy prescribed for greater than 12 hours per day) or nocturnal oxygen.
* Other Disease Abnormalities: Historical or current evidence of clinically significant or rapidly progressing or unstable cardiovascular, neurological, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the analysis if the disease/condition exacerbated during the study; Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures, or unable to continue their current COPD medications.
* Alcohol and Drug Abuse: A known or suspected history of alcohol or drug abuse within the last 2 years.
* A history of hypersensitivity to any components of the study inhaler (e.g., lactose, magnesium stearate). In addition, patients with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Prior or Ongoing use of the ELLIPTA inhaler (including both investigational and commercially available product).
* Investigational Product: Subjects who have received an investigational drug and/or medical device within 30 days of entry into this study (Screening/Visit 1), or within five drug half-lives of the investigational drug, whichever is longer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-10-01; Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were naive to ELLIPTA (trade name of dry powder inhaler owned by GlaxoSmithKline) inhaler use and had an established diagnosis of Chronic Obstructive Pulmonary Disease (COPD) participated in this study.
Groups:
- Placebo ELLIPTA Inhaler: Participants received study placebo via ELLIPTA inhaler at Visit 1 (Day 1) for use with their current daily inhaled COPD medication(s) that were to be continued during the study. Participants were instructed to take one inhalation from the ELLIPTA inhaler once daily at the same time each day until Day 28. At Visit 2 (Day 28), participants completed Version A or B of the ELLIPTA Inhaler Questionnaire as per randomisation.
Period: Overall Study
Arm/Group | Placebo ELLIPTA Inhaler
Started | 278
Completed | 266
Not Completed | 12
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Placebo ELLIPTA Inhaler
Number analyzed (Participants) | 278
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 147
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 28
  American Indian or Alaskan Native | 1
  White-White/Caucasian/European Heritage | 249

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With COPD Who Rate the Use of the ELLIPTA Inhaler as Easy or Very Easy, Among Those Who Demonstrate Correct Use of the Inhaler at the End of the Study.
Description: Participants rated how easy it was to use the ELLIPTA inhaler, using a four-point Likert scale (1-very easy, 2-easy, 3-difficult, 4-very difficult). "Easy to use" was defined as the combination of an "easy" or "very easy" rating choice. The percentage was reported overall for the single treatment group along with a 95% confidence interval (CI) for the percentage calculated using the exact binomial distribution. The percentage is based off the number of participants analyzed i.e the number of subjects in the MITT population (subjects who received a dose of study medication and were randomised).
Time Frame: Day 30
Population: Modified Intent-to-Treat (mITT) Population: all participants who were screened and received at least one dose of study treatment (placebo) and were randomised to receive the ELLIPTA inhaler ease of use questionnaire version A or B at Visit 2. Only participants with data available at the analysis time point were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo ELLIPTA Inhaler
Number analyzed (Participants) | 266
Percentage | 93 [90 to 96]

2. Secondary Outcome: The Percentage of Participants Who Rated the Ability to Tell How Many Doses Were Remaining in the ELLIPTA Inhaler as Easy or Very Easy at the End of the Study.
Description: Participants rated how easy it was to determine how many doses were left in the ELLIPTA inhaler, using a four-point Likert scale (1-very easy, 2-easy, 3-difficult, 4-very difficult). "Easy to use" was defined as the combination of an "easy" or "very easy" rating choice. The percentage was reported overall for the single treatment group along with a 95% CI for the percentage calculated using the exact binomial distribution.
Time Frame: Day 30
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo ELLIPTA Inhaler
Number analyzed (Participants) | 266
Percentage of Participants | 99 [97 to 100]

3. Secondary Outcome: The Percentage of Participants Who Demonstrated Correct Use of the ELLIPTA Inhaler at the End of the Study.
Description: Participants' ability to correctly use the ELLIPTA inhaler was assessed at Visit 1 and Visit 2 using the Correct Use Checklist by an ELLIPTA trained health care professional. The percentage was reported overall for the single treatment group along with a 95% CI for the percentage calculated using the exact binomial distribution.
Time Frame: Day 30
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo ELLIPTA Inhaler
Number analyzed (Participants) | 266
Percentage of Participants | 97 [94 to 99]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of Visit 1 until completion of Visit 2 (up to Day 30)
Description: The analysis population used for SAEs and non-serious AEs was Intent-to-Treat population: all participants who were screened and received at least one dose of study treatment (placebo)
Arm/Group | Placebo ELLIPTA Inhaler
Serious Adverse Events (participants affected / at risk) | 4/278
Other Adverse Events (participants affected / at risk) | 0/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo ELLIPTA Inhaler (N=278)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.